CLINICAL TRIAL: NCT00522574
Title: A Phase 1 Dose-Escalation Study of the Safety, Pharmacokinetics, and Pharmacodynamics of XL019 Administered to Subjects With Myelofibrosis
Brief Title: A Safety Study of XL019 in Adults With Myelofibrosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to emerging safety data
Sponsor: Exelixis (Industry)
Responsible Party: Chunyan Song, MD/Senior Manager, Clinical Research, Exelixis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL019-001
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2011-04

CONDITIONS: Myeloproliferative Disorders; Myelofibrosis; Polycythemia Vera; Thrombocythemia, Essential
Keywords: Myeloproliferative Disorders
MeSH Terms: conditions — Myeloproliferative Disorders; Primary Myelofibrosis; Polycythemia Vera; Thrombocythemia, Essential

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: XL019 — gelatin capsules supplied in 5-mg, 25-mg, and 100-mg strengths

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of XL019 in adults with myelofibrosis. XL019 is a selective inhibitor of the cytoplasmic tyrosine kinase JAK2. JAK2 is activated by cytokine and growth factor receptors and phosphorylates members of the STAT family of inducible transcription factors. Activation of the JAK/STAT pathway promotes cell growth and survival, and is a common feature of human tumors. JAK2 is activated by mutation in the majority of patients with myelofibrosis, polycythemia vera and essential thrombocytosis and appears to drive the inappropriate growth of blood cells in these conditions.

ELIGIBILITY:
Inclusion Criteria:

* The subject has primary myelofibrosis (PMF), post-polycythemia vera MF, or post-essential thrombocythemia MF and requires therapy, including subjects who have received prior MF-directed therapy and relapsed or subjects with refractory disease; or if newly diagnosed, then with intermediate or high risk according to the Lille scoring system.
* The subject is unwilling to undergo or is not a candidate for peripheral stem cell/bone marrow transplant.
* The subject is ≥18 years old.
* The subject has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
* The subject has adequate organ function.
* The subject has the capability of understanding the informed consent document and has signed the informed consent document.
* Sexually active subjects (male and female) must use medically acceptable methods of contraception during the course of the study.
* Female subjects of childbearing potential must have a negative pregnancy test at screening.
* The subject has had no diagnosis of malignancy or evidence of other malignancy for 2 years prior to screening for this study (except non-melanoma skin cancer or in situ carcinoma of the cervix).

Exclusion Criteria:

* The subject has uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within 3 months, or cardiac arrhythmias.
* The subject is pregnant or breastfeeding.
* The subject is known to be positive for the human immunodeficiency virus (HIV).
* The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-08

PRIMARY OUTCOMES:
To evaluate the safety, tolerability, maximum tolerated dose, and dose-limiting toxicities of XL019 as a single agent when orally administered in subjects with PMF, post-PV MF, or post-ET MF. | Assessed at periodic visits

SECONDARY OUTCOMES:
Determine plasma pharmacokinetics, evaluate pharmacodynamic correlates, and estimate renal elimination of XL019 | Assessed at periodic visits
Evaluate preliminary efficacy of XL019 as a single agent when administered orally | Assessed at periodic visits

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - UCSF - Division of Hematology/Oncology, San Francisco, California
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mt. Sinai School of Medicine, New York, New York
  - MD Anderson Cancer Center, Houston, Texas